CLINICAL TRIAL: NCT00621452
Title: A Pilot Study to Evaluate the Safety and Feasibility of Cellular Immunotherapy Using Genetically Modified Autologous CD20-Specific T Cells For Patients With Relapsed or Refractory Mantle Cell and Indolent B Cell Lymphomas
Brief Title: Genetically Engineered Lymphocytes, Cyclophosphamide, and Aldesleukin in Treating Patients With Relapsed or Refractory Mantle Cell Lymphoma or Indolent B-Cell Non-Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2154.00; NCI-2010-00416 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2008-02-21; First posted 2008-02-22 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Nodal Marginal Zone B-cell Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Cyclophosphamide; aldesleukin; Interleukin-2; Polymerase Chain Reaction; Gene Rearrangement; Sentinel Lymph Node Biopsy; Flow Cytometry; Enzyme-Linked Immunosorbent Assay

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (autologous CD20 specific T-cells) (Experimental): CHEMOTHERAPY: Patients receive cyclophosphamide IV over 60 minutes.
  IMMUNOTHERAPY: Beginning 2 days after completion of cyclophosphamide, patients receive autologous CD20-specific T-cells IV over 30 minutes. Treatment repeats every 2-5 days for 3 courses.
  MAINTENANCE THERAPY: Beginning 2 hours after the last T-cell infusion, patients receive low-dose aldesleukin subcutaneously twice daily for 14 days.
  Subjects who have achieved at least a partial remission lasting a minimum of 6 months may, on a case-by-case basis, receive additional stored T cells following relapse.
  Interventions: Biological: therapeutic autologous lymphocytes; Drug: cyclophosphamide; Biological: aldesleukin; Genetic: polymerase chain reaction; Genetic: gene rearrangement analysis; Procedure: lymph node biopsy; Biological: genetically engineered lymphocyte therapy; Procedure: bone marrow aspiration; Other: flow cytometry; Other: laboratory biomarker analysis; Other: enzyme-linked immunosorbent assay

INTERVENTIONS:
Biological: therapeutic autologous lymphocytes — Given IV
  Other Names: AL; Autologous Lymphocytes; autologous T cells
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: aldesleukin — Given subcutaneously
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Genetic: polymerase chain reaction — Correlative studies
  Other Names: PCR
Genetic: gene rearrangement analysis — Correlative studies
Procedure: lymph node biopsy — Optional correlative studies
  Other Names: Biopsy of Lymph Node
Biological: genetically engineered lymphocyte therapy — Receive genetically modified T cells
Procedure: bone marrow aspiration — Optional correlative studies
Other: flow cytometry — Correlative studies
Other: laboratory biomarker analysis — Correlative studies
Other: enzyme-linked immunosorbent assay — Correlative studies
  Other Names: ELISA

SUMMARY:
This phase I trial is studying the side effects of giving genetically engineered lymphocytes together with cyclophosphamide and aldesleukin in treating patients with relapsed or refractory mantle cell lymphoma or indolent B-cell non-Hodgkin lymphoma. Placing a gene that has been created in the laboratory into white blood cells may make the body build an immune response to kill cancer cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Aldesleukin may stimulate the white blood cells to kill lymphoma cells. Giving genetically engineered lymphocytes together with cyclophosphamide and aldesleukin may be an effective treatment for mantle cell lymphoma and B-cell non-Hodgkin lymphoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility, safety and toxicity of cellular immunotherapy utilizing ex-vivo expanded autologous T cells genetically modified to express a "second generation' cluster of differentiation (CD)20-specific scFvFc:CD28:CD137:zeda chimeric immunoreceptor in patients with recurrent or refractory CD20+ mantle cell or indolent lymphoma.

SECONDARY OBJECTIVES:

I. To determine the duration of in vivo persistence of adoptively transferred CD20-specific T cells transfected with a CD20-specific scFvFc:CD28:CD137:zeda chimeric immunoreceptor.

II. To assess the trafficking of CD20-specific T cells to lymphoma masses. III. To evaluate the development of host anti-CD20 scFvFc:CD28:CD137:zeda chimeric immunoreceptor and anti-neomycin-resistance gene (NeoR) immune responses in study subjects.

OUTLINE:

CHEMOTHERAPY: Patients receive cyclophosphamide IV over 60 minutes.

IMMUNOTHERAPY: Beginning 2 days after completion of cyclophosphamide, patients receive autologous CD20-specific T-cells IV over 30 minutes. Treatment repeats every 2-5 days for 3 courses.

MAINTENANCE THERAPY: Beginning 2 hours after the last T-cell infusion, patients receive low-dose aldesleukin subcutaneously twice daily for 14 days.

Treatment continues in the absence of disease progression or unacceptable toxicity.

Subjects who have achieved at least a partial remission lasting a minimum of 6 months may, on a case-by-case basis, receive additional stored T cells following relapse.

After completion of study treatment, patients are followed up weekly for one month, monthly for 1 year, and then annually for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects with immuno histopathologically documented CD20+ mantle cell lymphoma, follicular non-Hodgkin lymphoma (NHL), small lymphocytic lymphoma/chronic lymphocytic leukemia, marginal zone, or lymphoplasmacytic NHL of any age, gender, or ethnic group who have relapsed or are refractory to conventional chemotherapy and who are not eligible for Fred Hutchinson Cancer Research Center (FHCRC)/University of Washington Medical Center (UWMC) transplant protocols (or who refuse participation in transplant protocols)
* Willingness to sign an informed consent and undergo study tests
* Willingness to receive cytoreductive chemotherapy, if necessary to debulk tumors prior to T cell administration, and to receive cyclophosphamide for lymphodepletion
* Serologic evidence of prior exposure to Epstein-Barr virus (EBV)
* Meets safety criteria to undergo leukapheresis
* Hemoglobin > 9.0 gm/dL
* White blood cell (WBC) > 2500 per microliter
* Alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x Upper Limit of Normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x Upper Limit of Normal
* Creatinine =< 1.6 mg/dL
* Willingness to use acceptable (barrier or hormonal methods) birth control as appropriate during the course of the study

Exclusion Criteria:

* Treatment with fludarabine or cladribine within the previous 2 years prior to apheresis
* Known central nervous system involvement with NHL
* Pulmonary involvement with NHL; a diagnosis of pulmonary lymphoma will be based in part on findings from chest computed tomography (CT) and, if clinically appropriate, lung biopsy
* Exposure to chemotherapeutic agents (standard or experimental) or other immunosuppressive therapies less than four weeks prior to apheresis; patients must have recovered from acute side effects of such therapy
* Positive serology for human immunodeficiency virus (HIV)
* Active Hepatitis B or Hepatitis C infection
* History of hypersensitivity reactions to murine proteins or seropositivity for human anti-mouse antibody (HAMA)
* Requirement for corticosteroid therapy during the study period unless used specifically for amelioration of toxicity induced by transferred cells
* Treatment with anti-CD20 antibodies (rituximab, tositumomab, ibritumomab) within 4 months prior to start of T cell infusions
* Patients with lymph nodes in excess of 5 cm in diameter at time of T cell infusion
* Patients with > 5000 circulating CD20+ lymphocytes per mm^3 at time of T cell infusion
* Previous allogeneic stem cell transplantation
* Life expectancy less than 90 days
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-08; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Feasibility of transfecting and expanding the necessary numbers of T cells and the types of problems and toxicities which might be encountered, graded according the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0 | Up to 2 years after final T cell infusion
  A true grade 3 or higher toxicity rate in excess of 20% attributed to T cell infusions will be considered grounds for stopping the study and amending the protocol to lower the cell infusion doses. If there ever exists sufficient evidence to suggest that the true T cell-related toxicity rate (grade 3 or higher, with the exception of fever > 40 degrees Celsius lasting less than 24 hours) exceeds 20%, the study will be stopped.

SECONDARY OUTCOMES:
Comparison of the percentages of CD20-specific T cells and malignant B cells present in the blood before and after each T cell infusion | Up to 4 weeks after the third infusion
  Numbers and percentages of CD20-specific T cells and of malignant B cells will also be quantified in lymph node (LN) and bone marrow (BM).
Immune response as assessed by ELISA and percent chromium release in cytotoxicity assays | Up to 12 months following treatment
  Means, medians and standard deviation (S.D.) of the Ab titers observed will be computed.
Absolute numbers of T cells expressing the chimeric T Cell receptor (cTCR) per cubic uL of blood | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian Till, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

REFERENCES:
- [Derived] Till BG, Jensen MC, Wang J, Qian X, Gopal AK, Maloney DG, Lindgren CG, Lin Y, Pagel JM, Budde LE, Raubitschek A, Forman SJ, Greenberg PD, Riddell SR, Press OW. CD20-specific adoptive immunotherapy for lymphoma using a chimeric antigen receptor with both CD28 and 4-1BB domains: pilot clinical trial results. Blood. 2012 Apr 26;119(17):3940-50. doi: 10.1182/blood-2011-10-387969. Epub 2012 Feb 3. PMID 22308288